CLINICAL TRIAL: NCT06876896
Title: Comparative Study of Intra-abdominal Pressure Using Accuryn Monitoring System During Pulsed Field Ablation (PFA) for Treatment of Atrial Fibrillation and/or Atrial Flutter Under Sedation.
Brief Title: Intra-abdominal Pressure (IAP) During PFA Treatment of A-fib/ A-Flutter
Acronym: IAP
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Wake Forest University Health Sciences (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: IRB00124904
Record Dates: First submitted 2025-03-10; First posted 2025-03-14 (Actual); Last update posted 2025-12-17 (Actual); Status verified 2025-12

CONDITIONS: Intra-Abdominal Hypertension
Keywords: Atrial Fibrillation; Atrial Flutter; Pulsed Field Ablation
MeSH Terms: conditions — Intra-Abdominal Hypertension; Atrial Fibrillation; Atrial Flutter

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- Accuryn Foley catheter placement (Experimental): foley catheter is made to measure intra-abdominal pressure
  Interventions: Device: Accuryn Foley catheter device

INTERVENTIONS:
Device: Accuryn Foley catheter device — Accuryn foley catheter placed on all subjects after consent who are having treatment for atrial flutter or atrial fibrillation

SUMMARY:
The purpose of this study is to investigate the intra-abdominal pressure utilizing the Accuryn monitoring system during pulsed field ablation procedures in the electrophysiology lab compared to the type of anesthetic utilized.

DETAILED DESCRIPTION:
Intra-abdominal pressure (IAP) may play a role in patient outcomes during ablation procedures, as increased IAP could indicate potential adverse events. Such adverse events include aspiration of stomach contents, which can lead to respiratory issues post procedure and unplanned admission to the hospital post procedure. Potrero Medical has manufactured a foley based monitoring system that has been FDA cleared for the indication of measuring intra-abdominal pressure. The Accuryn monitor allows for continuous, real-time measurement of IAP and urine output, providing data that may enhance procedural safety and provide insights into any physiological responses unique to Pulsed Field Ablation (PFA). This study aims to compare PFA in terms of safety, efficacy, and IAP changes based on type of anesthesia received.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients receiving pulse field ablation procedures for standard of care treatment of atrial fibrillation and/or atrial flutter.
* Eligible for Foley catheter placement with no contraindications to Intra-abdominal pressure (IAP) monitoring.

Exclusion Criteria:

* Patients under the age of 18 will be excluded.
* History of intra-abdominal surgery within the past 6 months.
* Known contraindications to bladder catheterization or catheter ablation; history of prostate issues / Benign prostatic hyperplasia (BPH) or frequent urinary tract infections
* Pregnant or breastfeeding individuals
* History of chronic obstructive pulmonary disease (COPD) with home oxygen use

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2026-03 (Estimated); Primary Completion 2026-06-30 (Estimated); Study Completion 2026-07-30 (Estimated)

PRIMARY OUTCOMES:
Intra-abdominal pressure under Pulsed Field Ablation (PFA) under general anesthesia | hour 2
  intra-abdominal pressure during PFA when general anesthetic is utilized
Intra-abdominal pressure under Pulsed Field Ablation (PFA) under sedation | hour 2
  intra-abdominal pressure during PFA when anesthesia is sedation

SECONDARY OUTCOMES:
Incidence of Hiccups | hour 2
  incidence of hiccups occurring during the planned procedure
Amount oral secretions | hour 2
  Amount of oral secretions
Number of post-operative intubations | hour 2
  Number of incidences requiring postoperative intubation after procedure
Total urine output | hour 2
  Total urine output
Number of urinary tract infections | day 7
  Number of urinary tract infections in the week postoperatively
Number of unplanned admissions to the hospital | hour 2
  Number of unplanned admissions to the hospital

CONTACTS AND LOCATIONS:
Overall Officials: Karuna Rajkumar, MD, Principal Investigator — Wake Forest University Health Sciences
Locations (1):
- Wake Forest Health Sciences, Winston-Salem, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No